CLINICAL TRIAL: NCT01025973
Title: A New Approach by Mass Spectrometry for Evaluation and Validation of New Biomarkers of Fetus and Mother
Brief Title: Evaluation and Validation of New Biomarkers by Mass Spectrometry
Acronym: DG7
Status: Completed | Type: Observational
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Jean-Luc Ardilouze, Endocrinologist, researcher, Université de Sherbrooke
Other Study IDs: 09-110
Record Dates: First submitted 2009-12-03; First posted 2009-12-04 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine, whole blood, cord blood, plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diabetes Mellitus: Patients with type 1, type 2 or gestational diabetes mellitus
- Normal pregnancy: Patient without diabetes mellitus

SUMMARY:
The investigators will perform biochemical and metabolic evaluations on cord blood, venous blood of the mother and urine of the foetus and mother using time-of-flight and tandem mass spectrometry. The investigators could evaluate, dose and validate gestational diabetes mellitus biomarkers of the fetus and mother.

ELIGIBILITY:
Inclusion Criteria:

For women:

* Aged 18 or more
* 24 weeks of gestation or more
* Type 1, type 2 or gestational diabetes mellitus for group 1
* Without diabetes for group 2.

For newborn:

* 37 weeks of gestation or more
* Birth weight 2500 g or more

Exclusion Criteria:

* Multiple birth

Min Age: 1 Day | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Women with or without diabetes and their newborn.
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2009-10; Primary Completion 2011-05 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Foetal HbA1c | At delivery

SECONDARY OUTCOMES:
Foetal acetylated Hb | At delivery

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc Ardilouze, MD, PhD, Principal Investigator — Université de Sherbrooke
Locations (1):
- Centre de recherche clinique Etienne-Le Bel du CHUS, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dupont FO, Hivert MF, Allard C, Menard J, Perron P, Bouchard L, Robitaille J, Pasquier JC, Auray-Blais C, Ardilouze JL. Glycation of fetal hemoglobin reflects hyperglycemia exposure in utero. Diabetes Care. 2014 Oct;37(10):2830-3. doi: 10.2337/dc14-0549. Epub 2014 Jul 10. PMID 25011951